CLINICAL TRIAL: NCT03834038
Title: Prospective, Open-label Trial to Evaluate Efficacy of Lyophilized Fecal Microbiota Transplantation for Treatment of Recurrent C. Difficile Infection
Brief Title: Lyophilized Fecal Microbiota Transplantation for Recurrent Clostridioides Difficile Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Christine Lee, MD, Vancouver Island Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDI.LYO.FMT; NCT02592343 (obsolete NCT alias)
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Lyophilized Fecal Microbiota Transplantation (Experimental): Eligible participants with history of recurrent or refractory CDI
  Interventions: Drug: Lyophilized Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Lyophilized Fecal Microbiota Transplantation — Lyophilized FMT

SUMMARY:
The primary goal is to study participants with recurrent C. difficile infection (CDI) treated with lyophilized fecal microbiota transplantation (FMT). The safety, clinical response and relapse rate in patients will be assessed.

DETAILED DESCRIPTION:
Recurrence of CDI following a course of standard antibiotic therapy is high, especially in the elderly patients over 65 years of age, in hospitalized and in the immunocompromised patients. As CDI is characterized by intestinal dysbiosis. Fecal Microbiology Transplantation (FMT) has been investigated as alternative treatment for CDI and has been determined to be effective and safe. One of the major challenges of offering FMT is the availability of suitable donors. A donor may no longer be able to continue to donate for a number of reasons and this may lead to temporary interruption of FMT in centers which offer the program. In order to continue to offer FMT whenever needed, we will investigate the efficacy of lyophilized FMT. The lyophilization (freeze-drying) process works by dehydrating a frozen donor stool sample to complete dryness, using controlled temperature and pressure gradients. This lyophilized process results in a powdered form of the sample. Studies have shown that lyophilized donor stool samples have similar microbial compositions as the same fresh sample.The technique of freeze drying has been used for decades for the industrial storage of microbes and has been used. Preliminary study of lyophilized stool for FMT has been performed in dogs. Preliminary efficacy data in dogs with inflammatory bowel disease suggest equal efficacy as compared to fresh stool, although controlled study has yet to be performed. Should the lyophilized FMT (L-FMT) demonstrate to be equally or more effective than frozen FMT, there would be significant advantages. As with frozen FMT, lyophilized FMT will allow patients to receive FMT immediately as it can take up to two weeks for a donor's screening laboratory testing results to be available. Lyophilized FMT will also be more cost effective as less number of donors will need to be screened given the prolonged shelf life of lyophilized FMT which can be kept at above the freezing temperature. 9 This will also allow wider distribution and accessibility especially to the regions with limited capacity to manufacture FMT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years or older.
* Able to provide informed consent.
* Willing and able to comply with all the required study procedures.
* A positive stool test for C. difficile toxin/gene using either PCR or enzyme immunoassay within 3 months of recruitment unless patient taking treatment specifically for CDI for more than 3 months.
* History of at least ≥ 2 recurrent CDI where recurrence is deﬁned as return of diarrhea consistent with CDI within 8 weeks following CDI symptom resolution for at least 24 hours after a minimum of 10-day course of standard antibiotic therapy for each episode and/or ongoing symptoms consistent with CDI* (defined below) despite at least 7 days of treatment using oral vancomycin at a minimum dose of 250 mg four times daily.

  * Symptoms of CDI include: diarrhea deﬁned as: 3 or more unformed bowel movements in 24 hours for a minimum of 2 days with no other causes for diarrhea

Exclusion Criteria:

* Planned or actively taking another investigational product
* CDI symptom-free for 3 or more weeks following completion of CDI treatment
* Patients with neutropenia with absolute neutrophil count <0.5 x 109/L
* Evidence of toxic megacolon or gastrointestinal perforation on abdominal x-ray
* Active gastroenteritis due to Salmonella, Shigella, shiga toxin-producing E. coli, Yersinia or Campylobacter.
* Presence of colostomy
* Unable to tolerate FMT or enema for any reason.
* Requiring systemic antibiotic therapy for more than 7 days.
* Actively taking Saccharomyces boulardii or other probiotic; yogurt is allowed
* Severe underlying disease such that the patient is not expected to survive for at least 30 days.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, Principal Investigator — Vancouver Island Health Authority
Locations (1):
- Vancouver Island Health Authority, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants must have laboratory or pathology-confirmed diagnosis of recurrent CDI based on Society for Healthcare epidemiology of America SHEA definition, recurrence defined as return of diarrhea and positive stool test after period of symptom resolution within 8 weeks of the first episode and has received at least 10-day oral course of Vancomycin
  Eligible participants at time of screening will discontinue antibiotic 24-48 hours prior to scheduled FMT
Groups:
- Open Label Lyophilized Fecal Microbiota Transplantation: Open label for eligible participants with history of recurrent or refractory CDI
  Evaluate treatment efficacy as determined by no recurrence of CDI-related diarrhea at 13 weeks after receiving up to 2 lyophilized FMTs without the need for an intervention (antibiotics or frozen or lyophilized FMT as per investigator's decision) specifically for recurrence of CDI.
Period: Overall Study
Arm/Group | Open Label Lyophilized Fecal Microbiota Transplantation
Started | 158
Completion of 2-year Follow-up | 132
Completed | 132
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Lyophilized Fecal Microbiota Transplantation
Number analyzed (Participants) | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.25 (17.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: No Recurrence of CDI-related Diarrhea at 13 Weeks From Last LYO-FMT
Description: No recurrence of CDI-related diarrhea at 13 weeks following last FMT without the need for an intervention antibiotics or additional FMT specifically for CDI recurrence.
Time Frame: 13 weeks from last FMT
Population: 140 included in per-protocol analysis for primary endpoint 18 excluded as died/withdrew before week 13
Measure: Number; unit: participants
Groups:
- Open Label Lyophilized Fecal Microbiota Transplantation: Eligible participants treated with LYO-FMT
  Evaluate treatment efficacy as determined by no recurrence of CDI-related diarrhea at 13 weeks after receiving up to 2 lyophilized FMTs without the need for an intervention (antibiotics or frozen or lyophilized FMT as per investigator's decision) specifically for recurrence of CDI.
Arm/Group | Open Label Lyophilized Fecal Microbiota Transplantation
Number analyzed (Participants) | 140
participants | 106

ADVERSE EVENTS:
Time Frame: 1 year 2 months
Arm/Group | Open Label Lyophilized Fecal Microbiota Transplantation
All-Cause Mortality (participants affected / at risk) | 10/158
Serious Adverse Events (participants affected / at risk) | 14/158
Other Adverse Events (participants affected / at risk) | 15/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Lyophilized Fecal Microbiota Transplantation (N=158)
Cardiac event (Cardiac disorders) | 4 (4) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Genitourinary dysfunction (Renal and urinary disorders) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term,
C. difficile infection (Infections and infestations) | 3 (3)
leukocytosis (Blood and lymphatic system disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term,
Falls (Injury, poisoning and procedural complications) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term,
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term,
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Lyophilized Fecal Microbiota Transplantation (N=158)
Common Non-Serious (Gastrointestinal disorders) | 15 (15) — 10% constipation 10% increased flatulence 8% abdominal pain

LIMITATIONS AND CAVEATS:
One of the significant limitations of the study was the open-labelled nature of the study and the introduction of inherent bias but attempts were made to reduce the outcome bias by tracking the consistency and the number of bowel movements during the 13-week follow-up period; the stool was tested for CD toxin/gene when the participants experienced symptoms consistent with recurrent CDI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT03834038/Prot_SAP_000.pdf